CLINICAL TRIAL: NCT06645197
Title: A Multicenter, Single-Arm, Open-Label, IIT Clinical Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of a Single Intrathecal Injection of SNUG01 in Patients with Amyotrophic Lateral Sclerosis (ALS)
Brief Title: An IIT Clinical Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of a Single Intrathecal Injection of SNUG01 in Patients with Amyotrophic Lateral Sclerosis
Acronym: ALS
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: SineuGene Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Fan Dongsheng, Professor, Chief Physician, Peking University Third Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTP-SNUG01-IIT-02
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Gene therapy; AAV (adeno-associated virus); ALS; Neuromuscular Diseases; Motor Neuron Disease; Nervous System Diseases
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuromuscular Diseases; Motor Neuron Disease; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3 single Ascending Dose Levels (Experimental): The study will be open-label with an initial plan to explore 3 dose levels of SNUG01 in approximately 7 to 10 Participants in total. Each Participant will receive a single dose of SNUG01 delivered via intrathecal (IT) infusion and will be followed for up to 5 years after administration.
  Interventions: Drug: SNUG01

INTERVENTIONS:
Drug: SNUG01 — Recombinant adeno-associated virus serotype 9 capsid containing human SG001 expression cassette

SUMMARY:
This is a multicenter, open-label, single-arm investigator-initiated clinical study designed to evaluate the safety, tolerability, and preliminary efficacy of SNUG01 in patients with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
SNUG01 is a gene therapy designed to deliver a protective protein gene to the central nervous system. Safety will be the primary focus during the initial 24 weeks post-treatment (primary study period). After the primary study period, participants will be assessed for both safety and efficacy for up to a total of 5 years following SNUG01 treatment.

ELIGIBILITY:
Inclusion Criteria:

1.Able to understand and voluntarily sign the informed consent form, the informed consent form must be signed before performing any clinical trail procedures.

2.18~80 years old (including 18 and 80 years old), both male and female. 3.Must have been diagnosed with clinically probable ALS, clinically possible laboratory-supported ALS, or clinically definite ALS according to the revised version of the El Escorial World Federation of Neurology criteria.

4.Less than or equal to 36 months (inclusive) after the onset of symptoms of amyotrophic lateral sclerosis.

5.Body Mass Index (BMI) ≥19 kg/m2. 6.The forced vital capacity (FVC) in the screening period is greater than or equal to 70% of the estimated vital capacity.

7.Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) score ≥ 26 during the screening period, with scores of ≥ 4 in the three respiratory items (dyspnea, orthopnea, and respiratory insufficiency) on the ALSFRS-R.

8. Adequate organ function: Hematological: Neutrophil count≥1.5 × 10⁹/L, platelet count≥ 100 × 10⁹/L, Hemoglobin ≥90 g/L. Renal: Creatinine ≤1.5×ULN or creatinine clearance (CCr) ≥50 ml/min using the Cockcroft-Gault formula.

Hepatic: Total bilirubin (TBIL), alanine aminotransferase (ALT), aspartate aminotransferase (AST)≤2 × ULN, alkaline phosphatase (ALP) ≤ 3 × ULN.

Coagulation: International Normalized Ratio (INR), Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) ≤1.5 × ULN.

9.Subjects are not currently receiving riluzole or have been receiving a stable dose of riluzole for at least 4 weeks prior to the screening visit. Subjects treated with riluzole are expected to remain on the same dose throughout the study period.

9.Subjects are not currently treated with edaravone or are being treated with the approved standard regimen of edaravone. Subjects being treated with edaravone must have completed at least 1 cycle of treatment prior to the Screening Visit and are expected to continue treatment with edaravone throughout the study period.

10.Women of childbearing age must have a negative blood pregnancy test during the screening period and be non-lactating. Female subjects of childbearing age (women of childbearing age include premenopausal women and women within 2 years after menopause, except those who have undergone bilateral tubal ligation, complete oophorectomy or hysterectomy.) and male subjects whose partners are women of childbearing age must Agree to use effective contraceptive methods throughout the study period, such as abstinence, double barrier contraceptive methods, condoms, intrauterine devices and other non-drug contraceptive measures, and are not allowed to donate sperm or eggs.

Exclusion Criteria:

1. Serum anti-AAV9 neutralizing antibody (Nab) titer > 1:100 at the time of screening.
2. There are contraindications to lumbar puncture during the screening period (including but not limited to skin infection at the administration site and signs or symptoms of increased intracranial pressure), receiving any active intrathecal therapy, and having implants for drainage of cerebrospinal fluid (CSF). Inserted shunt, presence of implanted central nervous system (CNS) cannula, or any condition that prevents CSF collection.
3. There are other diseases related to motor neuron dysfunction (progressive bulbar palsy, primary lateral sclerosis, cervical spondylosis, lumbar spondylosis, etc., idiopathic inflammatory myopathy), which may confuse or cover up the diagnosis of ALS.
4. Previously required invasive ventilation or tracheotomy due to ALS disease, or currently using non-invasive ventilation support with an average of ≥16 hours/day.
5. Previous history of gene therapy, hematopoietic stem cell transplantation, and solid organ transplantation.
6. The patient has poorly controlled acute or chronic respiratory diseases, including but not limited to: chronic obstructive pulmonary disease, severe asthma, severe pneumonia, active tuberculosis.
7. Those who have been implanted or the researchers estimate that they will need to implant a diaphragmatic pacing system during the study period.
8. Any thromboembolic events occurred within 6 months before the first administration, such as deep vein thrombosis, pulmonary arteriovenous embolism, jugular vein embolism, etc..
9. Received another drug for the treatment of ALS disease (including but not limited to sodium phenylbutyrate (PB), taurine diol (TURSO), tauroursodeoxycholic acid (TUDCA) within 4 weeks before the first dose ) or ursodeoxycholic acid (UDCA), biologics, etc. except riluzole and edaravone).
10. Autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathies, mixed connective tissue disease, overlap syndrome, etc.) within 30 days prior to the Screening Period, or ongoing immune-related therapy (e.g., corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin, rituximab, leflunomide, hydroxychloroquine, interleukin 2 antagonists, etc.), except for intranasal, inhaled, ocular, topical topical, intra-articular corticosteroid therapy, or physiologic replacement therapy with corticosteroids.
11. Suffering from active or uncontrolled infection (including but not limited to: infectious pneumonia, sepsis, herpes zoster infection) within 4 weeks before the first administration, or chronic bacterial infection that is considered unacceptable according to the investigator's judgment ( medical history such as tuberculosis).
12. Have undergone major surgery within 4 weeks before the first administration, or have not recovered from previous treatment-related adverse events (AE) to ≤ grade 1 (CTCAE 5.0), except alopecia.
13. Participated in another clinical study within 4 weeks before the first administration, unless it is an observational (non-intervention) clinical study.
14. Any febrile illness occurred within 14 days before the first administration.
15. Have been vaccinated within 14 days before the first dose.
16. Patients with poorly controlled hypertension (refers to resting blood pressure after treatment: systolic blood pressure (SBP) > 160 mmHg or diastolic blood pressure (DBP) > 100 mmHg).
17. Arterial oxygen saturation and/or finger pulse oxygen saturation <93% after treatment with oxygen therapy or noninvasive respiratory support (<16 hrs/day) at the time of screening, as determined by the investigator.
18. Hypersensitivity to prednisolone, other glucocorticoids or their excipients.
19. Positive hepatitis B surface antigen (HBsAg) or positive hepatitis B core antibody (anti-HBcAb) with peripheral blood HBV DNA titer ≥ 1.0E+02 IU/mL.; positive hepatitis C virus (HCV) antibody with positive HCV RNA results; positive human immunodeficiency virus (HIV) antibody; or positive treponemal antibody for syphilis.
20. The following cardiovascular and cerebrovascular diseases, including but not limited to:

    QTc interval (corrected using Fridericia formula) average value: males QTc > 450 ms, females QTc > 470 ms.

    Echocardiogram showing left ventricular ejection fraction (LVEF) < 50% or below the lower limit of normal (whichever is higher).

    History of heart failure of class III-IV (NYHA classification). Myocardial infarction, unstable angina, poorly controlled arrhythmia, cerebrovascular accident or transient ischemic attack occurred within 6 months before the first administration;
21. Mental illness that may affect compliance with the test requirements: unstable mental illness, cognitive dysfunction, dementia or alcohol dependence, etc.
22. Other conditions that the researcher thinks are not suitable for participating in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2024-10-16 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2029-10-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ascending doses of intrathecally administered SNUG01 in Participants with ALS | Each visit in 1 year after administration
  Safety and tolerability, including adverse events (AE), vital signs, physical examination, clinical laboratory tests (hematology, blood chemistry, urinalysis, coagulation, cardiac enzymes, etc.) and 12 electrocardiograms,etc.

SECONDARY OUTCOMES:
Characterization of Immune Response to SNUG01 | up to 1 years
  Development of ADAs (antidrug antibodies) and neutralizing antibodies of SNUG01 and AAV9 in blood and cerebrospinal fluid ( CSF )
Characterization of the Effect of intrathecally administered SNUG01 | 3 months, 6months
  Change from Baseline in the Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R), the Rasch-Built Overall Amyotrophic Lateral Sclerosis Disability Scale（ROADS）and the Amyotrophic Lateral Sclerosis Assessment Questionnaire 40 (ALSAQ 40) total scores to Month 3 and Month 6
Characterization of the Effect of intrathecally administered SNUG01 | 3 months, 6 months,12 months
  The Change from baseline in forced vital capacity (FVC) to month 3, month 6 and month 12
Characterization of the Effect of intrathecally administered SNUG01 | 3 months, 6 months,12 months
  The change from baseline in Medical Research Council (MRC) on M3, M6 and M12 after IT administration of SNUG01.
Evaluate the long-term safety and tolerability of intrathecally administered SNUG01 in Participants with ALS | up to 5 years
  Number of participants with treatment-related adverse events and serious adverse events,including vital signs, physical examination, clinical laboratory tests (hematology, blood chemistry, urinalysis, coagulation, cardiac enzymes, etc.) and 12 electrocardiograms,etc.

OTHER OUTCOMES:
To evaluate the viral shedding after SNUG01 treatment | Up to 5 years
  Monitor the viral shedding in blood, saliva, urine, and feces
To explore the potential biomarkers in ALS subjects | 6 months, 12 months
  The change in the levels of SG001 protein , neurofilament light chain (NfL), interferon-γ (IFN-γ) in CSF and Blood after treatment of SNUG01

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fujian, Fuzhou
  - JiangSu Provincce Hospital, Nanjing, Jiangsu
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No